CLINICAL TRIAL: NCT01136122
Title: Effects of Positive Airway Pressure (PAP) Treatment of Obstructive Sleep Apnea (OSA) in Patients With Heart Failure
Brief Title: Effects of PAP Treatment of OSA in Patients With Heart Failure
Acronym: OSA-MRI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Ulysses Magalang MD (Other)
Responsible Party: Sponsor-Investigator, Ulysses Magalang MD, Medical Director, Sleep Medicine-East, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2009H0304
Record Dates: First submitted 2010-05-17; First posted 2010-06-03 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2016-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CPAP Arm (Active Comparator): Receive effective CPAP treatment for one month
  Interventions: Device: CPAP Treatment
- Control Arm (No Intervention): Receive no treatment for one month

INTERVENTIONS:
Device: CPAP Treatment — Effective CPAP treatment for one month
  Other Names: CPAP
  Arms: CPAP Arm

SUMMARY:
The purpose of this study is to see if treatment of OSA with the CPAP device makes a difference to insulin resistance and heart disease.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) has been seen frequently in persons who develop insulin resistance and heart disease. Insulin resistance is a condition in which the body produces insulin but does not use it properly. Insulin helps the body use glucose for energy. Insulin resistance increases the chance of developing type II diabetes and heart disease.

One method of treatment for OSA is with continuous positive airway pressure (CPAP). This treatment is given by a device named CPAP. There are many different types of CPAPs available on the market that are FDA approved.

The purpose of this study is to see if treatment of OSA with the CPAP device makes a difference to insulin resistance and heart disease. This study will measure insulin resistance by testing the glucose level in the blood, and testing the levels of special protein found in blood, that are known to increase the sensitivity to insulin and decrease progression of heart disease. The heart disease will be measured by cardiac MRI. Glucose testing and cardiac MRI's are normal testing procedures for people who have OSA and heart disease, however will be conducted more frequently than normal and therefore are for research purposes. The specialized blood testing is for research purposes only.

ELIGIBILITY:
Inclusion Criteria:

* 18 and < 75 years of age.
* Apnea-hypopnea index (AHI) of at least 15/hr based on overnight polysomnography.
* New York Heart Association Class 3 or less.
* LV ejection fraction <45% based on a prior imaging study (as measured within one year of baseline studies).
* Absence of exacerbation of heart failure requiring hospitalization within the previous 3 mos.
* Optimal pharmacologic therapy at the highest tolerated dose [3].

Exclusion Criteria:

* Use of anti-diabetic medications
* Primary valvular heart disease
* Unstable angina
* Myocardial infarction, cardiac surgery, or revascularization procedure within the previous 3 months
* Uncontrolled hypertension defined as systolic blood pressure >160 mm Hg or diastolic blood pressure >100 mm Hg.
* Active smoking (Patient should not have smoked for at least 1 month prior to baseline studies and has the intention not to smoke for the duration of the study period)
* Use of illicit drugs
* Current use of home oxygen therapy
* Requirement for a bi-level machine to treat sleep apnea
* Use of corticosteroids
* Creatinine clearance < 30ml/min (calculated from serum creatinine)
* Pregnant women will be excluded as pregnancy interferes with glucose and adiponectin. Additionally the contrast used in the cardiac MRIs may be harmful to unborn babies. Females of child bearing potential must agree to use effective contraception during the trial.
* Any contraindication to CMR (Cardiovascular magnetic resonance) imaging such as ferromagnetic foreign body, orbital metal, cerebral aneurysm clip, pacemaker, defibrillator, neurostimulator, allergy to gadolinium-based contrast, or severe claustrophobia. The standard FDA and OSUMC's screening guidelines for MRI safety will be followed.
* Inability or unwillingness to provide consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Increase in circulating levels of adiponectin (Ad) and/or high-molecular-weight (HMW) Ad. | One month

SECONDARY OUTCOMES:
Increased levels of Ad and/or HMW Ad associate with improvements in insulin sensitivity and heart function in patients with known left ventricular (LV) systolic dysfunction. | One month

CONTACTS AND LOCATIONS:
Overall Officials: Ulysses Magalang, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No